CLINICAL TRIAL: NCT02899013
Title: Description of Perianal Lesions in a Cohort of Crohn's Disease Patients
Acronym: LAPCROHN
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LAPCROHN
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Crohn Disease
Keywords: Perianal Lesions
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — Observational study to describe Perianal Lesions in a Cohort of Crohn's Disease Patients.

SUMMARY:
The perianal lesions (LAP) specific for Crohn's disease have been reported in 1938, six years after the first cases of luminal disease. If phenotypic data of the latter are well documented today, those of perianal disease remain inadequately described. The reasons are numerous: understated symptoms by patients, elementary semiotics proctology ignored by practitioners, lack of validated classifications to track these violations and challenges to undertake clinical trials to high standard of proof in view of these variables, etc. ... Moreover, the impact of these LAP varies across studies (10-80%). in addition to the above-mentioned reasons, these results are also due to the different definitions of LAP used in the studies, their collection in reference centers versus tertiary centers, their potential occurrence at any time of disease progression, their greater frequency in case of distal disease (12% for infringement isolated ileal, 15% in breach ileo colic, 41% in case of colonic involvement and 91% in case of rectal involvement). Yet the specific LAP should be better documented because they are a factor of poor prognosis of Crohn's disease.

DETAILED DESCRIPTION:
The perianal lesions (LAP) specific for Crohn's disease have been reported in 1938, six years after the first cases of luminal disease. If phenotypic data of the latter are well documented today, those of perianal disease remain inadequately described. The reasons are numerous: understated symptoms by patients, elementary semiotics proctology ignored by practitioners, lack of validated classifications to track these violations and challenges to undertake clinical trials to high standard of proof in view of these variables, etc. ... Moreover, the impact of these LAP varies across studies (10-80%). in addition to the above-mentioned reasons, these results are also due to the different definitions of LAP used in the studies, their collection in reference centers versus tertiary centers, their potential occurrence at any time of disease progression, their greater frequency in case of distal disease (12% for infringement isolated ileal, 15% in breach ileo colic, 41% in case of colonic involvement and 91% in case of rectal involvement). Yet the specific LAP should be better documented because they are a factor of poor prognosis of Crohn's disease.

In practice, Crohn's disease specific LAP are described in the UFS Cardiff classification. She is currently the most used even if the inter-observer reproducibility has never been demonstrated. This is an anatomical and pathophysiological classification distinguishes two types of LAP: primary, specific lesions (cracks and ulcers), and secondary lesions, consequences of mechanical complications (strictures) or infectious (fistulas and abscesses) lesions primary. The cracks are often multiple, broad and deep base and may occur in any quadrant of the anus. They may be painless and are not usually associated with sphincter hypertension. They constitute 20 to 35% of the LAP. Ulcerations realize profound substance of losses, based on an inflammatory tissue banks and have loosened, edematous. They often focus on the sub-pectineal portion of the anal canal and have an extension in height and depth. They are rarer: 5 to 10% of LAP. Stenoses are either functional, due to sphincter spasm and then reversible or organic, short or long fibrous membrane and irreversible. They usually occur after healing of ductal ulcers or abscesses. They represent 35% of the LAP. Fistulas may be secondary to infection of an anal gland Hermann and Desfosses or complicate a crack or anorectal ulcer. These are the most common LAP: 50 to 70%.

The epidemiology of non-specific LAP, ie "non-primary" and "no side", in Crohn's disease patients is even more unclear. However, the management of these lesions in patients at high risk of incontinence and for whom quality of life is affected by their chronic disease should be subject to special precautions. Prevalence of hemorrhoidal disease, estimated at 7% in a recent study, so is probably undervalued. The conservative therapeutic approach is consensus even though some recent studies have shown no complications after hemorrhoidectomy in patients with quiescent disease. Crohn's disease patients also have an excess risk poorly quantified develop various skin lesions anoperineal: secondary lesions to chronic diarrhea, fungal infections, contact dermatitis, paradoxical reactions to anti-TNF, autoimmune diseases associated, etc ... Finally, the effect of immunosuppression on the risk of anal cancer in Crohn's disease patients (with or without LAP) is not clearly known. Several authors have demonstrated an excess risk of infections Papillomavirus and intraepithelial neoplastic lesions of the anus in transplant treated with azathioprine and there is a risk of degeneration in severe injuries, and old chronicles. Monitoring could therefore be necessary in these sub-immune suppressor patients in the long term but there are currently no recommendations.

In short, the specific LAP or not Crohn's disease are poorly understood although their presence worsens the quality of life of patients and in some cases, is a factor of poor prognosis luminal disease. The purpose of this study is to describe the set of LAP (including specific or non-inflammatory disease lesions) in a cohort of patients with Crohn's disease.

Study Objectives

* accurately describe the LAP primary, secondary and "non-primary, not secondary" Crohn's patient cohort and obtain data including:

  * The type of injury
  * Their proportion
  * The treatment they have already been
  * Their impact on anal continence
  * Their impact on quality of life
  * Their field occurrence
  * The phenotypic profile of the associated luminal disease.
* establish a possible causal link between certain lesions and certain treatments.
* identify some injuries possibly worse prognosis.

Methodology

* non-interventional study
* prospective cohort.
* multicenter recruitment.
* Data collection in two steps:

  * In consultation:

    * initials, sex and patient age
    * phone
    * tobaccological profile
    * potential obstetric and surgical history
    * intestinal transit (across Bristol)
    * Data from the proctology examination (nonspecific lesions and classification UFS Cardiff)
    * activity profile of specific LAP (PDAI score Irvine)
    * impact of LAP on anal incontinence (Wexner score)
    * phenotypic profile of the luminal disease (classification of Montreal)
    * activity profile of luminal disease (Harvey-Bradshaw Index)
    * impact on quality of life (GIQLI the questionnaire)
    * previous treatments, current or proposed amendment if, Crohn's disease and LAP
    * serum CRP.
  * By phone, if necessary, in a second time to complete any missing data.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosed, all confused phenotype
* Perianal reached whatever its phenotype (specific or non-Crohn's disease).

Exclusion Criteria:

* Refusal or inability of the patient to be eventually reached by telephone
* Psychiatric pathology and / or non-understanding of the French language making the collection of random data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease diagnosed patients, all confused phenotype
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of PDAI Score | Day 15
  activity profile of specific LAP (PDAI score of Irvine)

SECONDARY OUTCOMES:
Assessment of Wexner score | Day 15
  impact of LAP on anal incontinence (Wexner score)
Assessment of phenotypic profile of the luminal disease (classification of Montreal) | Day 15
  Assessment of phenotypic profile of the luminal disease (classification of Montreal)
Assessment of Harvey-Bradshaw Index | Day 15
  activity profile of luminal disease (Harvey-Bradshaw Index)
Assessment of quality of life by GIQLI questionary | Day 15
  impact on quality of life (GIQLI questionary)

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided